CLINICAL TRIAL: NCT02264860
Title: Cohort 2: Researching Alveolar Macrophage Improvements With Supplements in HIV
Brief Title: Researching Alveolar Macrophage Improvements With Supplements in HIV
Acronym: RAISe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David M. Guidot, MD, Director, Division of Pulmonary, Allergy, & Critical Care Medicine, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00062730a; 1R01HL125042-01 (NIH)
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Zinc; S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nutritional Supplements Zinc and SAMe (Other): All men subjects will be started on 30 mg/day and women will be started on 25mg of elemental zinc plus 1600 mg/day of SAMe.
  Interventions: Dietary Supplement: Zinc and SAMe

INTERVENTIONS:
Dietary Supplement: Zinc and SAMe — The subjects will have the supplements dispensed at visit 2. They will be contacted weekly for the next three weeks to ensure that they are tolerating the supplements without significant side-effects. If these side-effects are significant then the dose of zinc will be decreased for all subjects to 15 mg of elemental zinc/day; if symptoms persist the SAMe dose will then be decreased by 25% (to 1200 mg/day) and then by 50% (to 800 mg/day) if necessary until the supplements are tolerated. 12 mg of zinc and 800 mg of SAMe is the lowest dose possible.

SUMMARY:
HIV infection causes systemic zinc deficiency and oxidative stress that impairs host immunity in the alveolar space.The purpose of this study is to see if taking two nutritional supplements, zinc and SAMe (S-adenosylmethionine), can improve lung health and immune function in persons with HIV.

The investigators hypothesize that long-term dietary supplementation with zinc and the glutathione precursor SAMe will enhance pulmonary host immune function in HIV-infected individuals who do not respond adequately to ART alone.

DETAILED DESCRIPTION:
This new proposal entitled "The alveolar macrophage pool is a reservoir of HIV" addresses a fundamental question; specifically, does the alveolar macrophage pool serve as a reservoir of HIV even when peripheral viral suppression is achieved by anti-retroviral therapy (ART) and if so, how does this reservoir alter the environment within the alveolar space and impair alveolar macrophage immune function? This is a critical question to address as lung infections remain the leading cause of death in persons living with HIV even when they are adherent to ART. There is compelling experimental evidence that HIV infection inhibits anti-oxidant defenses within the alveolar space and causes severe redox stress. Based on preliminary data presented in this proposal, the investigators hypothesize that HIV inhibits the expression and actions of Nrf2, the master transcription factor that activates the anti-oxidant response element (ARE), in part by inducing zinc deficiency in this vulnerable microenvironment, and thereby prevents the alveolar epithelium and the alveolar macrophage from generating glutathione and other anti-oxidants that are critically required to maintain a healthy redox potential within the alveolar space. The investigators further hypothesize that as a result of this targeted inhibition of the Nrf2-ARE signaling pathway, HIV promotes its own ability to infect alveolar macrophages and accumulate a large pool of intracellular pro-virus that produces a large HIV reservoir within the alveolar space. In parallel, HIV-induced oxidative stress shifts the alveolar macrophage toward alternative activation (so called 'M2 phenotype'). As a consequence, the innate immune capacity of the alveolar macrophage is impaired and this not only confers further resistance to clearing the viral reservoir but also renders the infected individual susceptible to serious lung infections. The investigators will leverage ongoing collaborative clinical studies in HIV-infected individuals. As a result, investigators not only have ongoing access to alveolar epithelial lining fluid and macrophages from well-defined subsets of HIV-infected individuals, they also have the expertise to apply state-of-the-art basic techniques in HIV pathogenesis, metabolomics, and redox signaling to test hypotheses. In parallel, the investigators are already conducting a prospective clinical trial of dietary zinc and S-adenosylmethionine (a thiol anti-oxidant that among its many actions increases the glutathione pool in the alveolar space) in HIV-infected individuals with inadequate immunological responses to ART (NCT01806870). This unique cohort will form the foundation for a greatly expanded clinical trial that will allow the investigators to test the corollary hypothesis that therapeutic strategies designed to improve zinc bioavailability and the redox potential within the alveolar space can enhance alveolar macrophage innate immune function and significantly decrease the HIV reservoir in the lung. This project will produce novel insights into how we can target the alveolar macrophage pool to decrease HIV burden as well as improve lung health in these vulnerable individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects living with HIV-1 infection who have been on anti-retroviral therapy (ART) for a minimum of 18 months and are followed longitudinally for their HIV healthcare in one of the study sites in Atlanta.
* Ability to give informed consent.

Exclusion Criteria:

* Documented history of cirrhosis or a direct bilirubin ≥ 2.0 mg/ld.
* Documentation of left ventricular ejection fraction < 40% or myocardial infarction within the past 6 months.
* End-stage renal disease requiring dialysis or a serum creatinine ≥ 2 mg/dL.
* Spirometry with Forced vital capacity (FVC) or Forced expiratory volume in 1 second (FEV1) < 70% of predicted value.
* Diabetes
* Known or possible pregnancy or attempting to become pregnant or breastfeeding
* BMI < 17
* Age < 21
* Parkinson's disease: these are all b/c the SAMe risks sections states that these pts will not qualify
* Bipolar disorder
* Bleeding disorders such as thrombocytopenia or significant gastrointestinal bleeding within the past year

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Dosage Efficacy | Three months
  Incidence of treatment-related adverse events, particularly gastrointestinal problems such as nausea, gastritis or diarrhea

SECONDARY OUTCOMES:
Change in exhaled breath condensate (EBC) levels of glutathione (GSH) | Baseline, 12 months
  Collection of exhaled breath condensate (EBC) is a non-invasive technique obtained by freezing and collecting exhaled breath that contains glutathione (GSH) from the lower airways. EBC GSH is measured is nmoles/µg urea.
Change in exhaled breath condensate (EBC) levels of glutathione (GSH) | Baseline, 24 months
  Collection of exhaled breath condensate (EBC) is a non-invasive technique obtained by freezing and collecting exhaled breath that contains glutathione (GSH) from the lower airways. EBC GSH is measured is nmoles/µg urea.

CONTACTS AND LOCATIONS:
Overall Officials: David M Guidot, MD, Principal Investigator — Emory University
Locations (1):
- Ponce De Leon Center, Atlanta, Georgia, United States

DOCUMENTS (1):
  • Informed Consent Form (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT02264860/ICF_000.pdf